CLINICAL TRIAL: NCT05035563
Title: Impact of an Early and Comprehensive Communication Strategy in the Prevention of Depressive Symptoms in Patients with Severe Covid-19, Their Families and Health Personnel
Brief Title: Impact of a Communication Strategy in the Prevention of Depressive Symptoms in Patients with Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Chile (Other); Universidad de La Frontera (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: COVID0921
Record Dates: First submitted 2021-03-27; First posted 2021-09-05 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2021-03

CONDITIONS: Critical Illness; Mechanical Ventilation; Covid19
Keywords: COVID-19; Depression post-ICU; Non-pharmacological intervention; Communication strategy
MeSH Terms: conditions — Critical Illness; COVID-19

STUDY DESIGN:
Intervention Model Description: Pre-intervention: The practices of each ICU will be maintained, until the moment that according to randomization corresponds to the beginning of the intervention, in each center
  Post-intervention: Integral and early strategy to facilitate communication between the family, patient and health team. For this it will be implemented written material, via the web (tablet and webmaster) and by telephone.
  It also includes strategies to support health teams, weekly multidisciplinary virtual meetings with the family, ICU diaries for family members.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional communication management (Pre-intervention) (No Intervention): Traditional communication practices are maintained, which consists of reporting the patient's medical conditions or specific requirements of the case, between the health team and the family.
  According to the social and administrative conditions of each centers, medical telephone information is provided on the conditions of the patients.
- Early and integral communication strategy (EICS) (Post-intervention) (Experimental): EICS that includes a bundle of various strategies that allow to favor communication and contact between family members, patients and health team.
  That considers the delivery of: (1) Receive timely and understandable information; (2) Receive visits, companionship, and spiritual assistance
  Interventions: Behavioral: Intervention. Early and integral communication strategy (EICS)

INTERVENTIONS:
Behavioral: Intervention. Early and integral communication strategy (EICS) — This intervention will be implemented in patients since they are hospitalized in the ICU where is expected:
  * Facilitate contact and communication between patients, families and the health team.
  * Respond to the communication needs of family members.
  * Reduce equipment overload and facilitate communication with families and patients, providing tools and timely support.
  * Build a positive and trusting relationship of relatives and patients with health teams.
  The intervention considers the following actions:
  1. - Training in communication to the health team
  2. - Written material
  3. - Family website
  4. - Standardized and daily telephone information
  5. - Health Team Support Strategy
  6. - Weekly multidisciplinary virtual meeting with the family
  7. - ICU diaries for family members
  Arms: Early and integral communication strategy (EICS) (Post-intervention)

SUMMARY:
The purpose of this study is to compare the effect of an early and integral communication strategy (EICS) versus standard care, on the rate of depressive symptoms at 3 months after discharge from the ICU, in patients with severe Covid-19, their family members and health personnel.

Evaluating the rate of depressive symptoms at 3 months after discharge from the ICU, with a) Hospital Anxiety and Depression, b) Posttraumatic Stress Disorder Checklist (S)

DETAILED DESCRIPTION:
We designed a pre-post intervention study, the groups were non-randomly allocated.

The study is implementation in 10 Chilean hospitals, admitting 350 patients.

Pre-intervention: The practices of each ICU will be maintained, until the moment that according to randomization corresponds the beginning of the intervention, in each center.

Post-intervention: EICS to facilitate communication between the family, patient and health team, through written material, via the web (tablet and webmaster) and by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years old
* Admitted to the ICU
* Requiring Mechanical Ventilation> 12 hrs due to COVID-19

Exclusion Criteria:

* Patients with therapeutic proportionality is defined early
* Patients with communication limitations (they do not speak Spanish) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of depressive symptoms | Third month post-discharge from ICU
  The rate of depressive symptoms after discharge from the ICU will be evaluated in patients with severe Covid-19, their relatives and health personnel with the instrument HADS (Hospital Anxiety and Depression Scale)

SECONDARY OUTCOMES:
Risk factors of depressive symptoms | Third month post-discharge from ICU
  Identify risk factors associated with depressive symptoms at 3 months post ICU in patients with severe Covid-19, their relatives and health team. Considering physical health, mental health and sociodemographic factors.
  To measure depressive symptoms will be used Hospital Anxiety and Depression Scale (HADS), total scores for depression range from 0 to 21, categorized as: normal (0-7), mild (8-10), moderate (11-14) or severe (15-21)
Functional independence post-ICU | Third month post-discharge from ICU
  Barthel will be used in patients, the score are ordered: 0-20 suggests total dependence, 21-60 severe dependence, 61-90 moderate dependence and 91-99 slight dependence, 100 independence
Functional independence post-ICU | Twelfth month post-discharge from ICU
  Barthel will be used in patients
Functionality Status post-ICU | Third month post-discharge from ICU
  Post-COVID-19 Functional Status (PCFS) will be used in patients, the score are : 0 = No functional limitations, 1=Negligible functional limitations, 2=Slight functional limitations, 3=Moderate functional limitations,4=Severe functional limitations, 5=death
Functionality Status post-ICU | Twelfth month post-discharge from ICU
  Post-COVID-19 Functional Status (PCFS) will be used in patients
Post traumatic stress post-ICU | Third month post-discharge from ICU
  This mental health condition will be evaluated in patients, family members and the health team, with the instrument Impact of Event Scale Revised (IES-R). Score Interpretation: 24-32: PTSD is a clinical concern, 33-38: This represents the best cutoff for a probable diagnosis of PTSD, 39 and above: This is high enough to suppress your immune system's functioning
Post traumatic stress post-ICU | Twelfth month post-discharge from ICU
  This mental health condition will be evaluated in patients, family members and the health team, with the instrument Impact of Event Scale Revised (IES-R).
Cognition status post-ICU | Third month post-discharge from ICU
  MOCA blind instrument will be applied to patients. The total possible score is 22 points; a score of 18 or above is considered normal
Cognition status post-ICU | Twelfth month post-discharge from ICU
  MOCA blind instrument will be applied to patients.
Quality of life post ICU | Third month post-discharge from ICU
  Euro Qol (EQ-5D) will be applied to patients. An EQ-5D summary index is derived by applying a formula that essentially attaches values (weights) to each of the levels in each dimension. The index can be calculated by deducting the appropriate weights from 1, the value for full health
Quality of life post ICU | Twelfth month post-discharge from ICU
  Euro Qol (EQ-5D) will be applied to patients.
ICU memories post ICU | Third month post-discharge from ICU
  ICU Memory Tool (ICUMT) will be applied to patients.In ICUMT, memories are categorized in subscales of factual memories, memories of feelings, and memories of delusion
ICU memories post ICU | Twelfth month post-discharge from ICU
  ICU Memory Tool (ICUMT) will be applied to patients.In ICUMT, memories are categorized in subscales of factual memories, memories of feelings, and memories of delusion
Anxiety post ICU | Third month post-discharge from ICU
  This mental health condition will be evaluated in patients, family members and the health team, with the instrument HADS total scores for anxiety range from 0 to 21, categorized as: normal (0-7), mild (8-10), moderate (11-14) or severe (15-21)
Anxiety post ICU | Twelfth month post-discharge from ICU
  This mental health condition will be evaluated in patients, family members and the health team
Rate of depressive symptoms | Twelfth month post-discharge from ICU
  The rate of depressive symptoms after discharge from the ICU will be evaluated in patients with severe Covid-19, their relatives and health personnel with the instrument HADS (Hospital Anxiety and Depression Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Alegria, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile - Medicina, Santiago, Santiago Metropolitan, Chile